CLINICAL TRIAL: NCT07170423
Title: Automated Text Message Reminders to Promote Hearing Aid Adoption
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Uchechukwu Megwalu, Professor of Otolaryngology - Head & Neck Surgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 82494
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Hearing Loss
Keywords: hearing loss; hearing aid; text message; patient reminders
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Automated Text Message Reminder (Experimental): Participants in the intervention group will receive automated text messages instructing them to obtain hearing aids. The messages will also include basic information on the prevalence and negative effects of hearing loss.
  Interventions: Behavioral: Automated text message reminder
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Automated text message reminder — Participants in the intervention group will receive automated text messages instructing them to obtain hearing aids. The messages will also include basic information on the prevalence and negative effects of hearing loss.
  Arms: Automated Text Message Reminder

SUMMARY:
Many individuals with hearing loss do not receive adequate hearing healthcare. Only about 30 percent of people that are found to have hearing loss during a hearing test go on to use hearing aids. The investigators propose to test the use of text message reminders to educate patients with hearing loss, and to encourage them to get hearing aids. The study objective is to examine whether automated text-messaging reminders increase the use of hearing aids among patients with hearing loss, who are hearing aid candidates.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adult patients who have been recommended for hearing aids.

Exclusion Criteria:

* Patients will be excluded if they use hearing aids or cochlear implants.
* Patients without a valid cellphone number will be excluded.
* Patients with dementia will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Likelihood of obtaining hearing aids | This outcome data will be collected 3, 6, 9, and 12 months after enrollment.
  Participants will be queried on whether they have obtained hearing aids since enrollment in the study. Participants who have not obtained hearing aids, will be asked to rate the likelihood that they would obtain hearing aids. Likelihood will be assessed on an 11-point visual analogue scale (VAS). Score range: 0 to 10 (0 = not likely, 10 = very likely). Participants who have already obtained hearing aids will be assigned a score of 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No